CLINICAL TRIAL: NCT05647876
Title: A Longitudinal Study to Identify Mechanisms of Menopause on Cardiovascular Disease Risk
Status: Recruiting | Type: Observational
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Lasse Gliemann, Associate Professor, University of Copenhagen
Other Study IDs: KISO STUDY
Record Dates: First submitted 2022-11-15; First posted 2022-12-13 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Menopause; Cardiovascular Diseases; Vascular Dilation; Physical Activity
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, muscle biopsy samples, urine samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
With the cessation of estrogen production at menopause, the risk of cardiovascular disease like arthrosclerosis, myocardial infarction and stroke increases dramatically. Physical activity is the single most powerful "drug" for maintaining and improving cardiovascular health, but recent data suggest that the positive effect of physical activity is lost at menopause. In this project the investigators will follow a cohort of 200 women from before the women enter menopause and until at least 10 years past menopause. By advanced invasive methodologies the investigators will monitor the changes that occur in the blood vessels of the circulation, the heart and the brain and combine this with microRNA sequencing of blood and tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Normal ECG
* Regular menstruation

Exclusion Criteria:

* Participation in other clinical projects
* Smokes or has smoked within the last 10 years
* On hormone therapy
* Has chronic diseases that are not expected, cf. the groups sought. Including heart problems, atrial fibrillation, cancer, immune diseases and previous strokes with functionally significant sequelae
* Being treated with oral steroids
* Has alcohol / drug abuse or is being treated with disulfiram (Antabus)
* Is unable to understand the contents of the document with informed consent or the experimental procedures
* Pregnancy or breastfeeding
* Systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg
* ovariectomy
* BMI>28

Ages: 40 Years to 61 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women between 40-61 years of age, who are menstruating regularly, but that are close to the menopause ( will be estimated through hormonal levels).
  It is anticipated that the population will have different physical activity levels, and the population will thus be stratified from this, to investigate the role of different habitual physical activity level.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2045-08 (Estimated)

PRIMARY OUTCOMES:
Invasive vascular function | pre, 1yr. 3yr. , 5 yr., 10 yr. and 20 yr. post menopause
  Changes in vascular function across the menopausal transition (pre, 1yr. 3yr. , 5 yr., 10 yr. and 20 yr. post menopause Vascular function is assessed by intra-arterial infusions of acetylcholine and epoprostenol) in the brachial artery using ultrasound doppler
Non-invasive vascular function | pre, 1yr. 3yr. , 5 yr., 10 yr. and 20 yr. post menopause
  Changes in vascular function across the menopausal transition (pre, 1yr. 3yr. , 5 yr., 10 yr. and 20 yr. post menopause Vascular function is assessed by flow-mediated dilation (FMD) in the brachial artery using ultrasound doppler

SECONDARY OUTCOMES:
Changes in skeletal muscle expression of protein | pre, 1yr. 3yr. , 5 yr., 10 yr. and 20 yr. post menopause
  Changes in skeletal muscle expression of protein across the menopausal transition, and with different physical activity levels. (pre, 1yr. 3yr. , 5 yr., 10 yr. and 20 yr. post menopause
  Western blots will be used to determine endothelial nitric oxide synthase (eNOS), cyclo-oxygenase 1 and 2, prostacyclin synthase, endothelin receptor A and B, VEGF (vascular endothelial growth factor), Thrombospondin-1, Flk-1 (VEGF receptor). All protein content measures will be presented as arbitrary units.
Changes in skeletal muscle and blood sample expression of RNA | pre, 1yr. 3yr. , 5 yr., 10 yr. and 20 yr. post menopause
  Changes in skeletal muscle and blood sample expression of RNA across the menopausal transition, and with different physical activity levels. (pre, 1yr. 3yr. , 5 yr., 10 yr. and 20 yr. post menopause.
  RNA sequencing will be used to determine changes in RNA profile, with specific focus on microRNA.
Blood pressure | pre, 1yr. 3yr. , 5 yr., 10 yr. and 20 yr. post menopause
  Changes in blood pressure across the menopausal transition

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Gliemann, PhD, Principal Investigator — Department of Nutrition, Exercise and Sports, University of Copenhagen, 2200 Copenhagen, Denmark
Locations (1):
- Deparment of Nutrition, Exercise and Sports, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No